CLINICAL TRIAL: NCT05088252
Title: Effects of Desflurane on the Quality of Anesthesia Recovery Period in Patients Undergoing Endonasal Endoscopic Pituitary Adenoma Resection#a Randomized Controlled Study
Brief Title: Desflurane and Anesthesia Recovery Period in Endonasal Endoscopic Pituitary Adenoma Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XUAN20211004
Record Dates: First submitted 2021-10-05; First posted 2021-10-21 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Pituitary Neoplasms
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane Inhalational Anesthesia (Experimental)
  Interventions: Drug: Desflurane
- Propofol Total Intravenous Anesthesia (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Desflurane — After induction, anesthesia will be maintained with 0.7-1.0 MAC desflurane and 0.05-0.3 μg/kg/min remifentanil.
  Arms: Desflurane Inhalational Anesthesia
Drug: Propofol — After induction, anesthesia will be maintained with 4-6mg/kg/h propofol and 0.05- 0.3 μg/kg/min remifentanil.
  Arms: Propofol Total Intravenous Anesthesia

SUMMARY:
Nasal packing is required after endoscopic pituitary adenoma resection. The patient can only breathe through the mouth. The blood and secretion in the nasal cavity may be inhaled into the trachea after the operation. GH-secreting pituitary adenoma causes pharyngeal soft tissue and tongue hypertrophy. These conditions increase the risk of respiratory obstruction and hypoxemia during anesthesia recovery. Propofol total intravenous anesthesia has a rapid effect and a low incidence of nausea and vomiting. Patients anesthetized with desflurane recover quickly is conducive to early recovery of respiratory function and orientation. This study intends to compare the effects of desflurane and propofol on the quality of anesthesia recovery period in patients undergoing endonasal endoscopic pituitary adenoma resection and to provide clinical evidence for the use of desflurane in neurosurgical anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years;
* Elective endoscopic transsphenoidal resection of pituitary adenomas;
* ASA status I-III;
* Informed consent signed by patients.

Exclusion Criteria:

* emergency surgery;
* complicated with cerebrovascular disease;
* complicated with pulmonary disease, oxygen saturation below 95% without oxygen;
* expected to retain endotracheal intubation;
* preoperative disturbance of consciousness was not compatible with assessment;
* complicated with primary hypothyroidism;
* previous history of cervical surgery, burns, and radiotherapy;
* BMI >30kg/m2;
* invasive pituitary adenoma with Knosp grade 4.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Time required of the Aldrete score reached 9 points after drug withdrawal. | immediately after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ruquan Han, Beijing, Beijing Municipality, China